CLINICAL TRIAL: NCT00146120
Title: Risk-Adapted Therapy of Acute Myeloid Leukemia of Adults (18-60 Years) According to the Cytogenetic Result
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Prof. Dr. Reinhard Marre, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLHD98A
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2008-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Etoposide

INTERVENTIONS:
Drug: Idarubicin
Drug: Cytosin-Arabinosid
Drug: Etoposide
Drug: All-trans Retinoid acid

SUMMARY:
The concept of the investigators risk-adapted multicenter treatment trial for younger adults, AML HD98A, is based on the results of the AML HD93 trial and on published data. Definition of risk groups is different compared to the AML HD93 trial; high-risk: refractory disease after first induction therapy and/or high risk karyotype [abn(3q), -5/5q-, -7/7q-, abn(12p), abn(17p), complex]; intermediate-risk: complete remission after induction therapy and intermediate risk karyotype [normal, abn(11q23), abn(16q22), other rare aberrations]; low-risk: complete remission after induction therapy and low risk karyotype [t(8;21)]. Patients exhibiting a t(15;17) were treated in a separated trial (APL HD95). Treatment consists of a first induction therapy with ICE followed by a second cycle ICE in case of response to first induction therapy. Patients with refractory disease after first induction therapy are assigned to a salvage therapy with A-HAM (all-trans retinoic acid, high-dose cytarabine and mitoxantrone) and the search for potential hematopoietic stem cell donors is extended from the family to unrelated persons. All patients achieving a CR after induction therapy with ICE are assigned to a first consolidation therapy with HAM. For intermediate-risk patients a peripheral stem cell or a bone marrow harvest are intended during the hematological recovery after the first consolidation. Second consolidation therapy was stratified according to the risk definition. For high risk patients a allogeneic transplantation is assigned from a related or unrelated donor preferentially after a dose-intensified conditioning therapy. All patients with intermediate risk and an HLA-matched family donor are assigned to allogeneic transplantation. Intermediate-risk patients without a family donor and normal karyotype at diagnosis are randomized between an autologous stem cell transplantation and a second course of HAM. The other intermediate-risk patients are assigned to autologous transplantation. For low-risk patients a second course of HAM is assigned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, de Novo or secondary after Myelodysplasy, or with therapy-induced AML after healed primary malignom; or refractory anemia with excess of blasts in transformation (RAEB-t); the diagnosis must be confirmed morphological, cytochemical and with immunological phenotyping
* Cytogenetical tests must be performed for each patient
* Age: 16 - 60 years
* All patients have to be informed about the character of the study. Written informed consent of each patient at study entry.

Exclusion Criteria:

* Organic insufficiency: Insufficiency of the kidneys (Crea > 1.5 x upper normal serum level), or insufficiency of the liver (bilirubin, SGOT or AP > 2 x upper normal serum level) uncaused by the AML; severe obstruction or restrictive ventilation disorder, heart failure with a ejection fraction < 0.5
* Secondary malignom
* Other severe diseases
* Pregnancy
* Participation in an concurrent clinical study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 1998-05; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
relapse-free survival | two years

SECONDARY OUTCOMES:
overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Döhner, Prof. Dr., Principal Investigator — University of Ulm
Locations (22):
- Austria (2):
  - Department of Hematology / Oncology, University Hospital of Innsbruck, Innsbruck
  - III Medical Department, Hematology and Oncology Center, Hanuschhospital Wien, Vienna
- Germany (20):
  - Department of General Internal Medicine, University Hospital of Bonn, Bonn
  - Department of Internal Medicine Hematology, Heinrich-Heine University, Düsseldorf
  - Department of Interial Medicine III, City Hospital Frankfurt Am Main - Höchst, Frankfurt
  - Medical Department IV, University of Gießen, Giessen
  - Department of Interial Medicine, Wilhelm-Anton-Hospital Goch, Goch
  - Centre of Interial Medicine, University of Göttingen, Göttingen
  - Medical Department III of Hematology and Oncology, General Hospital Altona, Hamburg
  - Department of Interial Medicine V, University of Heidelberg, Heidelberg
  - Department of Interial Medicine I, University Hospital of Saarland, Homburg
  - Medical Department II, City Hospital Karlsruhe gGmbH, Karlsruhe
  - Medical Department II, University Hospital of Kiel, Kiel
  - Department of Interial Medicine /Hematology and Oncology, Caritas Hospital Lebach, Lebach
  - I. Medical Department, City Hospital München-Schwabing, München
  - Medical Department III, Clinical Center rechts der Isar, München
  - Department of Hematology and Oncology, City Hospital Neunkirchen gGmbH, Neunkirchen
  - Department of Hematology and Oncology, Clinical Center of Oldenburg gGmbH, Oldenburg
  - Department of Hematologie and Oncology, Caritas Hospital St. Theresa Saarbrücken, Saarbrücken
  - Clinikal Cetner of Stuttgart, Center of Oncology, Stuttgart
  - Medical Department I, Clinical Center of Stuttgart, Stuttgart
  - Hospital of Barmherzige Brüder, I Medical Department, Trier

REFERENCES:
- [Derived] Prochazka KT, Pregartner G, Rucker FG, Heitzer E, Pabst G, Wolfler A, Zebisch A, Berghold A, Dohner K, Sill H. Clinical implications of subclonal TP53 mutations in acute myeloid leukemia. Haematologica. 2019 Mar;104(3):516-523. doi: 10.3324/haematol.2018.205013. Epub 2018 Oct 11. PMID 30309854
- [Derived] Papaemmanuil E, Gerstung M, Bullinger L, Gaidzik VI, Paschka P, Roberts ND, Potter NE, Heuser M, Thol F, Bolli N, Gundem G, Van Loo P, Martincorena I, Ganly P, Mudie L, McLaren S, O'Meara S, Raine K, Jones DR, Teague JW, Butler AP, Greaves MF, Ganser A, Dohner K, Schlenk RF, Dohner H, Campbell PJ. Genomic Classification and Prognosis in Acute Myeloid Leukemia. N Engl J Med. 2016 Jun 9;374(23):2209-2221. doi: 10.1056/NEJMoa1516192. PMID 27276561
- [Derived] Buchner T, Schlenk RF, Schaich M, Dohner K, Krahl R, Krauter J, Heil G, Krug U, Sauerland MC, Heinecke A, Spath D, Kramer M, Scholl S, Berdel WE, Hiddemann W, Hoelzer D, Hehlmann R, Hasford J, Hoffmann VS, Dohner H, Ehninger G, Ganser A, Niederwieser DW, Pfirrmann M. Acute Myeloid Leukemia (AML): different treatment strategies versus a common standard arm--combined prospective analysis by the German AML Intergroup. J Clin Oncol. 2012 Oct 10;30(29):3604-10. doi: 10.1200/JCO.2012.42.2907. Epub 2012 Sep 10. PMID 22965967
- [Derived] Gaidzik VI, Bullinger L, Schlenk RF, Zimmermann AS, Rock J, Paschka P, Corbacioglu A, Krauter J, Schlegelberger B, Ganser A, Spath D, Kundgen A, Schmidt-Wolf IG, Gotze K, Nachbaur D, Pfreundschuh M, Horst HA, Dohner H, Dohner K. RUNX1 mutations in acute myeloid leukemia: results from a comprehensive genetic and clinical analysis from the AML study group. J Clin Oncol. 2011 Apr 1;29(10):1364-72. doi: 10.1200/JCO.2010.30.7926. Epub 2011 Feb 22. PMID 21343560
- [Derived] Schlenk RF, Dohner K, Mack S, Stoppel M, Kiraly F, Gotze K, Hartmann F, Horst HA, Koller E, Petzer A, Grimminger W, Kobbe G, Glasmacher A, Salwender H, Kirchen H, Haase D, Kremers S, Matzdorff A, Benner A, Dohner H. Prospective evaluation of allogeneic hematopoietic stem-cell transplantation from matched related and matched unrelated donors in younger adults with high-risk acute myeloid leukemia: German-Austrian trial AMLHD98A. J Clin Oncol. 2010 Oct 20;28(30):4642-8. doi: 10.1200/JCO.2010.28.6856. Epub 2010 Aug 30. PMID 20805454
- [Derived] Kayser S, Schlenk RF, Londono MC, Breitenbuecher F, Wittke K, Du J, Groner S, Spath D, Krauter J, Ganser A, Dohner H, Fischer T, Dohner K; German-Austrian AML Study Group (AMLSG). Insertion of FLT3 internal tandem duplication in the tyrosine kinase domain-1 is associated with resistance to chemotherapy and inferior outcome. Blood. 2009 Sep 17;114(12):2386-92. doi: 10.1182/blood-2009-03-209999. Epub 2009 Jul 14. PMID 19602710